CLINICAL TRIAL: NCT07379749
Title: Impact of Positive Bile Cultures on Plastic Biliary Stent Exchange
Acronym: TEMPEST 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Colentina (Other)
Responsible Party: Principal Investigator, Andrei Voiosu, Lecturer Dr., Clinical Hospital Colentina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 42/12.12.2025
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Cholangitis
Keywords: early onset acute cholangitis after subsequent biliary stent occlusion

STUDY DESIGN:
Intervention Model Description: Patients with plastic biliary stent placement and a positive bile culture at index ERCP will be randomized into two groups: Group A, scheduled for early plastic stent exchange at 1 month, and Group B, scheduled for standard stent exchange at 3 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): standard follow up and stent exchange according to institutional norm
  Interventions: Other: stent exchange
- rapid exchange (Active Comparator): rapid call back in case of positive bile culture
  Interventions: Other: Scheduled biliary stent exchange at one month

INTERVENTIONS:
Other: stent exchange — standard stent exchange at three months according to the institutional norms
  Arms: Control
Other: Scheduled biliary stent exchange at one month — Patients within the active arm will have scheduled stent exchange at one month, in comparison to those in the control arm, which will have scheduled stent exchange at three months, according to the institutional norms in place
  Arms: rapid exchange

SUMMARY:
This prospective, unicenter, randomized controlled trial evaluates whether a positive bile culture at index ERCP with plastic stenting identifies patients who benefit from earlier stent exchange. Patients with no previous history of sphincterotomy and positive bile cultures after an ERCP will be randomized to stent exchange at 1 month versus 3 months to assess whether personalized scheduling reduces early stent occlusion and secondary acute cholangitis.

DETAILED DESCRIPTION:
A positive bile culture obtained at the index ERCP in patients with no previous history of sphincterotomy undergoing plastic biliary stenting may represent a key, yet currently largely ignored, predictor of early stent occlusion and subsequent acute cholangitis. Based on the findings of the TEMPEST Study, conducted in the Gastroenterology Department of Colentina Clinical Hospital (currently submitted for publication), which suggested a clinical benefit of earlier scheduled ERCP for stent exchange in this high-risk subgroup, we hypothesize that bile culture-guided scheduling of stent exchange can improve clinical outcomes.

To test this hypothesis, we propose a prospective, unicentric, randomized controlled trial comparing patients with positive bile cultures at index ERCP randomized to early stent exchange at 1 month versus standard exchange at 3 months. The primary objective is to determine whether personalized scheduling based on initial bile culture results reduces the incidence of early acute cholangitis, thereby offering a simple, low-cost strategy to optimize post-ERCP management and prevent further complications.

ELIGIBILITY:
Inclusion Criteria:

* All patients between 18 and 90 years old with native papilla and obstructive jaundice of any etiology requiring plastic biliary stent placement, with a positive bile culture at index ERCP who can provide written informed consent (obtained from the patient or legal caregiver).

Exclusion Criteria:

* prior ERCP attempts
* patients with bilio-digestive surgical or endoscopic anastomoses
* inability to provide informed consent due to cognitive, legal, or medical reasons
* scheduled surgical resection within one month after ERCP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Comparative analysis of the incidence rates of acute cholangitis in the scheduled stent exchange group, at one month, vs. standard stent exchange at three months | from enrollment to the end of treatment at three months
  The primary endpoint of this study is the incidence of cholangitis in patients with a positive bile culture at index ERCP with plastic stent placement. By comparing the outcomes between the 2 groups, the study aims to demonstrate that earlier stent exchange in this high-risk subgroup improves patient outcome by decreasing procedure-related complications, supporting a personalized management strategy instead of the current standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Colentina Clinical Hospital, Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No